CLINICAL TRIAL: NCT02016924
Title: A Phase 2/3, Multicenter, Open-label, Multicohort Study Evaluating Pharmacokinetics (PK), Safety, and Efficacy of Cobicistat-boosted Atazanavir (ATV/co) or Cobicistat-boosted Darunavir (DRV/co) and Emtricitabine/Tenofovir Alafenamide (F/TAF) in HIV-1 Infected, Virologically Suppressed Pediatric Participants
Brief Title: Study of Cobicistat-Boosted Atazanavir (ATV/co), Cobicistat-Boosted Darunavir (DRV/co) and Emtricitabine/Tenofovir Alafenamide (F/TAF) in Children With HIV
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-216-0128; 2013-001402-28 (EudraCT Number); IS000883 (Other: Argentina: The National Registry of Health Research (ReNIS))
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acquired Immune Deficiency Syndrome (AIDS); HIV Infections
Keywords: Pediatrics; Adolescents; HIV; HIV-1; Treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Atazanavir Sulfate; Darunavir; Cobicistat; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Part A and Part B (Experimental): Participants ages 12 to <18 years old will receive cobicistat 150 mg with either ATV or DRV plus background regimen (BR). The BR may contain additional antiretroviral agents except for the following disallowed agents: saquinavir, indinavir, nelfinavir, double protease inhibitor (PI) regimens, raltegravir, elvitegravir, efavirenz, nevirapine, delavirdine, maraviroc, etravirine, rilpivirine, dolutegravir, and investigational antiretroviral agents.
  Interventions: Drug: ATV; Drug: DRV; Drug: Cobicistat; Drug: BR
- Cohort 2 (Experimental): Participants aged 6 to <12 years old and ≥25 to <40kg will receive cobicistat 150 mg and F/TAF 200/25 mg with either ATV or DRV.
  Interventions: Drug: ATV; Drug: DRV; Drug: Cobicistat; Drug: F/TAF
- Cohort 3 (Experimental): Participants age ≥ 2 years old will receive cobicistat 90 mg and F/TAF 120/15 mg with either ATV or DRV.
  Interventions: Drug: ATV; Drug: DRV; Drug: Cobicistat; Drug: F/TAF
- Cohort 4 (Group 1) (Experimental): Participants age ≥ 4 weeks old weighing 14 to < 25 kg will receive cobicistat tablet for oral suspension (TOS) 90 mg, once daily and F/TAF TOS 120/15 mg, once daily with either ATV or DRV or lopinavir boosted by ritonavir (LPV/r). Minimum age and weight for ATV is ≥ 3 months and ≥ 5 kg, minimum age and weight for DRV is ≥ 3 years and ≥ 15 kg; participants receiving LPV/r will not receive cobicistat TOS.
  Interventions: Drug: ATV; Drug: DRV; Drug: LPV/r; Drug: Cobicistat TOS; Drug: F/TAF TOS
- Cohort 4 (Group 2) (Experimental): Participants age ≥ 4 weeks old weighing 10 to < 14 kg will receive cobicistat TOS 30 mg (twice daily) and F/TAF TOS 60/7.5 mg, once daily with either ATV or LPV/r. Minimum age and weight for ATV is ≥ 3 months and ≥ 5 kg, respectively; participants receiving LPV/r will not receive cobicistat TOS.
  Interventions: Drug: ATV; Drug: LPV/r; Drug: Cobicistat TOS; Drug: F/TAF TOS
- Cohort 4 (Group 3) (Experimental): Participants age ≥ 4 weeks old weighing 6 to < 10 kg will receive cobicistat TOS 30 mg (twice daily) and F/TAF TOS 30/3.75 mg, once daily with either ATV or LPV/r. Minimum age and weight for ATV is ≥ 3 months and ≥ 5 kg, respectively; participants receiving LPV/r will not receive cobicistat TOS.
  Interventions: Drug: ATV; Drug: LPV/r; Drug: Cobicistat TOS; Drug: F/TAF TOS
- Cohort 4 (Group 4) (Experimental): Participants age ≥ 4 weeks old weighing 3 to < 6 kg will receive cobicistat TOS 30 mg (twice daily) and F/TAF TOS 15/1.88 mg, once daily with either ATV or LPV/r. Minimum age and weight for ATV is ≥ 3 months and ≥ 5 kg, respectively; participants receiving LPV/r will not receive cobicistat TOS.
  Interventions: Drug: ATV; Drug: LPV/r; Drug: Cobicistat TOS; Drug: F/TAF TOS
- Cohort 5 (Group 1) (Experimental): Participants ages ≥ 4 weeks old weighing ≥ 10 to < 14 kg will receive F/TAF TOS 60/7.5 mg, once daily with the third unboosted drug.
  Interventions: Drug: Third Unboosted Drug; Drug: F/TAF TOS
- Cohort 5 (Group 2) (Experimental): Participants ages ≥ 4 weeks old weighing ≥ 6 to < 10 kg will receive F/TAF TOS 30/3.75 mg, once daily with the third unboosted drug.
  Interventions: Drug: Third Unboosted Drug; Drug: F/TAF TOS
- Cohort 5 (Group 3) (Experimental): Participants ages ≥ 4 weeks old weighing ≥ 3 to < 6 kg will receive F/TAF TOS 15/1.88 mg, once daily with the third unboosted drug.
  Interventions: Drug: Third Unboosted Drug; Drug: F/TAF TOS

INTERVENTIONS:
Drug: ATV — Capsules administered once daily according to dosing recommendations per product monograph
  Other Names: Reyataz®
  Arms: Cohort 1: Part A and Part B; Cohort 2; Cohort 3; Cohort 4 (Group 1); Cohort 4 (Group 2); Cohort 4 (Group 3); Cohort 4 (Group 4)
Drug: DRV — Tablets administered once daily according to dosing recommendations per product monograph
  Other Names: Prezista®
  Arms: Cohort 1: Part A and Part B; Cohort 2; Cohort 3; Cohort 4 (Group 1)
Drug: Cobicistat — Tablets administered orally once daily with food
  Other Names: GS-9350; Tybost®
  Arms: Cohort 1: Part A and Part B; Cohort 2; Cohort 3
Drug: BR — Background Regimen (BR) include Food and Drug Administration (FDA)-approved nucleos(t)ide reverse transcriptase inhibitors (NRTIs) including zidovudine (ZDV), stavudine (d4T), didanosine (ddI), abacavir (ABC), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), lamivudine (3TC), and emtricitabine (FTC).
  Arms: Cohort 1: Part A and Part B
Drug: F/TAF — Tablets administered orally once daily
  Other Names: Descovy®
  Arms: Cohort 2; Cohort 3
Drug: LPV/r — Solution administered orally
  Arms: Cohort 4 (Group 1); Cohort 4 (Group 2); Cohort 4 (Group 3); Cohort 4 (Group 4)
Drug: Third Unboosted Drug — ATV (administered orally), DRV (administered orally), and LPV/r (administered orally) would be general list but unspecified for sites.
  Arms: Cohort 5 (Group 1); Cohort 5 (Group 2); Cohort 5 (Group 3)
Drug: Cobicistat TOS — Tablets for oral suspension
  Other Names: GS-9350; Tybost®
  Arms: Cohort 4 (Group 1); Cohort 4 (Group 2); Cohort 4 (Group 3); Cohort 4 (Group 4)
Drug: F/TAF TOS — Tablets for oral suspension
  Other Names: Descovy®
  Arms: Cohort 4 (Group 1); Cohort 4 (Group 2); Cohort 4 (Group 3); Cohort 4 (Group 4); Cohort 5 (Group 1); Cohort 5 (Group 2); Cohort 5 (Group 3)

SUMMARY:
The goal of this clinical study is to learn more about the safety and dosing of study drugs, cobicistat-boosted Atazanavir (ATV/co), cobicistat-boosted darunavir (DRV/co) and emtricitabine/tenofovir alafenamide (F/TAF), in children (age ≥ 4 weeks to < 18 years) with HIV.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-1 infected, virologically suppressed males and females age ≥ 4 weeks to < 18 years (according to requirements of enrolling Cohort).
* Body weight at screening ≥ 25 to < 40 kg (Cohort 2); ≥ 14 to < 25 kg (Cohort 3); ≥ 3 to < 25 kg (Cohort 4); ≥ 3 to < 14 kg (Cohort 5).
* Stable antiretroviral (ARV) regimen for a minimum of 3 months prior to the screening visit.

  * Participants enrolled prior to implementation of Amendment 7: 2 nucleoside reverse transcriptase inhibitors (NRTIs) and ritonavir-boosted atazanavir (ATV/r) once daily or ritonavir-boosted darunavir (DRV/r) once daily or twice daily.
  * Participants enrolled after the implementation of Amendment 9:

    * Cohorts 2, 3 and 4 (Group 1): 2 NRTIs plus a third agent per local prescribing guidelines. Participants will switch from their current third agent to ATV or darunavir (DRV) at Day 1. Participants taking DRV must be on once-daily dosing or must switch to once daily at or prior to Day 1. Cohort 4 (Group 1), participants may also switch their current third agent to lopinavir boosted with ritonavir (LPV/r) at Day 1. Participants will switch their NRTI backbone to emtricitabine/tenofovir alafenamide (coformulated; Descovy®) (F/TAF).
    * Cohort 4 (Groups 2 to 4) and Cohort 5 (Groups 1 to 3): 2 NRTIs plus a third agent per local prescribing guidelines or treatment naive. Participants on treatment will switch from their current third agent to ATV or LPV/r (Cohort 4 (Groups 2 to 4)), or to a third unboosted agent (Cohort 5 (Groups 1 to 3)). Participants will switch their NRTI backbone to F/TAF.
* Participants undergoing dose modifications to their ARV regimen for growth or switching medication formulations are considered to be on a stable ARV regimen.
* Documented plasma human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) for ≥ 3 months preceding the screening visit:

  * Participants enrolled after the implementation of Amendment 9:

    * For Cohorts 2, 3, and 4 (Group 1), virologically suppressed ≥ 3 months preceding the screening visit: HIV-1 RNA < 50 copies/mL on a stable regimen (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL).
    * For Cohorts 4 (Groups 2 to 4) and Cohort 5 (Groups 1 to 3), on an ARV regimen irrespective of plasma HIV-1 RNA copies or treatment naive; a participant is considered treatment naive, if ARVs were given for prevention of mother-to-child transmission but not for HIV treatment.
  * For virologically suppressed participants, unconfirmed virologic elevations of HIV-1 RNA ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL (eg, < 20 copies/mL), the plasma HIV-1 RNA level cannot exceed 50 copies/mL on 2 consecutive HIV-1 RNA tests.
* Adequate renal function: Estimated glomerular filtration rate (eGFR) ≥ 90 mL/min/1.73m2 using the Schwartz formula. If ≥ 1 year old, eGFR greater than or equal to the minimum normal value for age using the Schwartz formula. If < 1 year old as follows:

  * Age minimum value for eGFR (mL/min/1.73 m2) > 28 days to ≤ 95 days is 30, ≥ 96 days to ≤ 6 months is 39, > 6 to < 12 months is 49.
* Participants must not have documented or suspected resistance to applicable study drugs including emtricitabine (Emtriva®) (FTC), TFV, ATV, DRV, or LPV. Participants < 14 kg (Cohorts 4 (Groups 2 to 4) and 5 (Groups 1 to 3)) with M184V/I AND HIV-1 RNA < 50 copies/mL will be allowed.
* Positive confirmatory HIV test (confirmatory nucleic acid-based testing if < 18 months of age).
* Cohort 4 (Groups 2 to 4) and Cohort 5 (Groups 1 to 3): Last dose of nevirapine or efavirenz, if applicable, ≥ 14 days prior to enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria do apply.

Ages: 4 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Parameter: AUCtau of ATV, DRV, TAF, and TFV | Predose on Day 1, and postdose up to Week 48
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
  AUCtau for ATV (Cohorts 1 Part A, 2, 3, and 4 [Groups 2 to 4]); DRV (Cohorts 1 Part A, 2, and 3); TAF (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 [Groups 1 to 3] taking F/TAF); and TFV (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 [Groups 1 to 3] taking F/TAF) will be reported.
Percentage of Participants Experiencing Treatment Emergent Adverse Events (AEs) Through Week 24 | First dose date up to Week 24 plus 30 days (Cumulative data through Week 24)
Percentage of Participants Experiencing Treatment Emergent Laboratory Abnormalities Through Week 24 | First dose date up to Week 24 plus 30 days (Cumulative data through Week 24)

SECONDARY OUTCOMES:
PK Parameter: Ctau of ATV, DRV, COBI, FTC and TFV | Predose on Day 1, and postdose up to Week 48
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
  Ctau for ATV (cohorts 1, 2, 3, and 4 (Groups 2 to 4)), DRV (cohorts 1, 2, and 3), COBI (except Cohort 5), FTC and TFV (cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
PK Parameter: Cmax of ATV, DRV, COBI, TAF, FTC and TFV | Predose on Day 1, and postdose up to Week 48
  Cmax is defined as the maximum observed concentration of drug.
  Cmax for ATV (Cohorts 1, 2, 3, and 4 [Groups 2 to 4]) and DRV (Cohorts 1, 2, and 3); for COBI (except Cohort 5); for TAF, FTC and TFV (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
PK Parameter: CL/F of ATV, DRV, COBI, TAF, FTC and TFV | Predose on Day 1, and postdose up to Week 48
  CL/F is defined as the apparent oral clearance following administration of the drug.
  CL/F for ATV (Cohorts 1, 2, 3, and 4 [Groups 2 to 4]) and DRV (Cohorts 1, 2, and 3); for COBI (except Cohort 5); for TAF, FTC and TFV (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
PK Parameter: Vz/F of COBI, TAF, FTC and TFV | Predose on Day 1, and postdose up to Week 48
  Vz/F is defined as the apparent volume of distribution of the drug.
  Vz/F for COBI (Except Cohort 5); for TAF (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF); for FTC and TFV (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
PK Parameter: AUCtau of COBI and FTC | Predose on Day 1, and postdose up to Week 48
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
  AUCtau for COBI (Except Cohort 5) and FTC will be reported.
PK Parameter: AUClast of TAF, FTC and TFV | Predose on Day 1, and postdose up to Week 48
  AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
  AUClast for TAF (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF); for FTC and TFV (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
PK Parameter: Clast of TAF | Predose on Day 1, and postdose up to Week 48
  Clast is defined as the the last observed quantifiable concentration of the drug in plasma.
  Clast for TAF (Cohorts 2, 3, 4 [Groups 1 to 4] and 5 taking F/TAF) will be reported.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to Week 48 plus 30 days (Cumulative data through Week 48)
Percentage of Participants Experiencing Clinically Significant Changes in Safety Laboratory Values | First dose date up to Week 48 plus 30 days (Cumulative data through Week 48)
Percentage of Participants with HIV-1 RNA < 50 Copies/mL at Week 24 and as Defined by the US FDA-defined Snapshot Algorithm | Week 24
Percentage of Participants with HIV-1 RNA < 50 Copies/mL at Week 48 and as Defined by the US FDA-defined Snapshot Algorithm | Week 48
Change from Baseline in CD4+ Cell Counts (cells/μL) at Week 24 | Baseline, Week 24
Change from Baseline in CD4+ Cell Counts (cells/μL) at Week 48 | Baseline, Week 48
Change from Baseline in Percentage of CD4+ Cells at Week 24 | Baseline, Week 24
Change from Baseline in Percentage of CD4+ Cells at Week 48 | Baseline, Week 48
Acceptability of COBI and F/TAF as Measured by Palatability Score | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (23):
- United States (7):
  - Pediatric Infectious Disease Associates, Long Beach, California
  - Peter Morton Medical Building, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - The George Washington University, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Health Science Center of Houston, Houston, Texas
- Argentina (2):
  - Hospital General de Agudos Cosme Argerich, Buenos Aires
  - Helios Salud, Buenos Aires
- South Africa (6):
  - University of the Free State, Bloemfontein
  - University of Stellenbosch, Cape Town
  - King Edward VIII Hospital, Durban
  - Rahima Clinical Trials, a Division of Wits Health Consortium (Pty) Ltd, Johannesburg
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria
  - Perinatal HIV Research Unit, Soweto
- Thailand (3):
  - HIV-NAT, Bangkok
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
- Uganda (3):
  - MU-JHU Research Collaboration/MU-JHU Care Ltd, Kampala
  - SICRA-TASO Mulago National Referral Hospital, Kampala
  - AMBSO Masaka Clinical Research Site, Masaka
- Imperial College Healthcare NHS Trust, London, United Kingdom
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-216-0128